CLINICAL TRIAL: NCT04117854
Title: Sunnaas International Network Pediatric Spinal Cord Injury Study - an International Multicenterstudy in Seven Countries
Brief Title: Spinal Cord Injury in the Pediatric Population - an International Multicenter Study
Acronym: SINpedSCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: Oslo Metropolitan University (Other); University of Oslo (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kirsti Skavberg Roaldsen, Professor, Sunnaas Rehabilitation Hospital
Other Study IDs: SINpedSCI2018
Record Dates: First submitted 2018-06-12; First posted 2019-10-07 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Pediatric ALL; Spinal Cord Injuries
Keywords: spinal cord injury; pediatric; qualitative interviews; web survey; international; multicenter; traumatic SCI; atraumatic SCI
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
INTRODUCTION: Due to the low incidence of pediatric spinal cord injury (SCI) and the high demand for knowledge and research, international cooperation is needed to build a solid and shared understanding of the extent of the problem, and also uniformity in treatment and measurement methods. The aim of the study is to map organization of care and rehabilitation of children and adolescents < 18 years of age with SCI, to explore qualitatively psychosocial aspects of individuals and to establish use of common outcome measures in 10 rehabilitation units from seven countries, cooperating within the Sunnaas International Network in Rehabilitation (SIN); China, USA, Russia, Israel, Palestine, Norway and Sweden.

METHOD: In Phase I two cross-sectional studies will be conducted to set the scene for the outcome studies following in Phase II (2020-2022). Phase I consists of a quantitative descriptive study using a websurvey to describe and compare the systems of care and delivery of inpatient rehabilitation services for pediatric SCI patients. In addition, a qualitative study will explore the psychosocial aspects of living with a childhood acquired SCI. Two adolescents, aged 13-17 years and at least 6 months post-acute treatment, from each unit will interviewed using a semi-structured interview guide. Ethical approval has been applied for in each unit, and the study is registered at ClinicalTrial-gov. A workshop for the 24 study team members, where the main focus was to ensure that data collection is conducted in a good manner, was held in May 2018, and data collection is expected finalized by 2020. Phase II (planning stage) will consist of methodological outcome studies.

DISCUSSION: Phase I of the study will broaden the body of knowledge on pediatric SCI internationally, thus enabling comparison, discussion and development of organizational models and quality of care and rehabilitation for young persons with SCI. Phase II will contribute to the use of common and reliable outcome measures for these patients.

DETAILED DESCRIPTION:
INTRODUCTION Spinal cord injury (SCI) before the age of 15 is rare affecting less than 1 in every 100 000 children. Over the past decade the management of pediatric spinal cord injury and the long-term outcomes have received increased attention, however, most research has its origin from the US. Thus, there is a need for more knowledge about occurrence and causes, functional recovery, activity, participation and quality of life in children and adolescents in other countries than the US. Moreover, a systematic review 2011 shows that there is limited evidence about the effectiveness of interventions for the management of children with SCI.

Knowledge regarding organization of care and rehabilitation is incomplete and differences between countries are substantial. Also, comparisons of data between countries and studies have been problematic due to differences in case definitions and age limits as to what is considered pediatric as opposed to adult SCI. Therefore, there is a need for international collaboration and research within the area of pediatric SCI with uniformity in methodology in the gathering of information and publication of the data to compare results between countries.

Due to the low incidence of pediatric SCI and the demand for more knowledge and research, international cooperation is needed for purposes of building a solid and common understanding of the scope of the problem and uniformity in management and methodology.

To reach this goal in the SIN context there is a need to benchmark between units, to highlight opportunities to improve systems of care and service delivery and to provide an understanding of the context of the units and the similarities and differences between them as this will be important for interpreting the results from subsequent phases of this project when patient outcomes are reported.

Exploration of psycho-social issues from the perspective of the affected young persons and their families will assist targeting issues that are clinically and socially relevant for future service and future research cooperation. In addition, to be able to gather information to compare results between countries it is important to establish use of common outcome measures.

AIMS AND OBJECTIVES Long term aim and objective The long-term goal of this research project is to optimize organization, care and rehabilitation in Norway and cooperating rehabilitation units internationally, to increase the awareness of subjective perceptions and psychosocial aspect of young persons with spinal cord injury, and to establish the use of outcome measures in local languages. Participants will be recruited from the rehabilitation hospitals cooperating within the Sunnaas International Network for Rehabilitation; Norway, Sweden, China, Russia, US, Israel, Palestine (SIN-units).

Specific aims and objectives

* To survey the SIN units in order to describe and compare the organization and delivery of inpatient rehabilitation services and systems of care for pediatric SCI patients
* To explore qualitatively psychosocial aspects of living with spinal cord injury in children and adolescents in SIN units using individual, semi-structured interviews

MATERIAL AND METHODS Study design This project is a cross sectional international multicenter study. A PhD-student is associated with the study (Oslo Metropolitan University/ Sunnaas Rehabilitation Hospital, start September 2019).

The first stage of the project (Phase I) will comprise a descriptive part (Study I, Web survey) and an explorative part (Study II, semi-structured interviews) conducted in clinical settings in Norway, Sweden, China, Russia, US, Israel and Palestine.

Recruitment The recruitment will be done within the units cooperating in the Sunnaas International Network for Rehabilitation (SIN).

The local principle investigator in each unit will be responsible for collecting data in Study I and recruiting individuals to participate in Study II of the study. Potentially eligible individuals with SCI will be identified from the departmental or institutional database. If no suitable database is present in an investigative site, recruitment through alternative databases will be explored and discussed with project collaborators.

Once identified, the study coordinator and local investigator will agree participant identification codes for the selected individuals. The study coordinator will allocate a three letter code (the first two letters will originate from the country of the study site, and the third from the name of the institution).

Inclusion criteria´s for the target group

* Children and adolescents (< 18 years)
* Diagnoses: either a non-traumatic or traumatic SCI after the age of 7
* Has been discharged from initial rehabilitation for 6 months or more

General Exclusion Criteria

• Diagnosis of severe neurological conditions affecting the cognition of the child or adolescent (e.g. as a result of encephalocele or acquired brain injury)

Participants Study I (descriptive study/ web survey). Ten rehabilitation units in Norway, Sweden, China, Russia, US, Israel and Palestine will be participating. The local principle investigator in each unit will be responsible for data collection.

Study II (explorative study/semi-structured interviews). Two individuals in each of the ten SIN units, fulfilling the inclusion criteria's, will be recruited. A maximum of 20 young informants 13-17 years will be interviewed and constitute the study group of the International qualitative study. In addition, all norwegian youth with SCI rehabilitated at Sunnaas Rehabilitation Hospital fulfilling the inclusion criteria and beeing13-17 years of age during the inclusion period, will be recruited and constitute the study group of the Norwegian qualitative study (6-10 persons). Pilot interviews will be conducted prior to data collection.

Data collection and analyzing Study I (descriptive study/ web survey) A web-survey based on clinical expertise and literature review have been developed in cooperation between Dr Peter W New, Spinal Rehabilitation Service, Caulfield Hospital, Australia and Norwegian clinicians and researchers with experience in pediatric SCI. The survey is a development and an adapted version of the survey used to conduct an international comparison of the organization of rehabilitation services and systems of care for adult patients with non-traumatic SCI in Italy, Ireland, India, Pakistan, Switzerland, the Netherlands, US, Australia and Canada.

The survey will be used to gather descriptive data to review the various forms of care and rehabilitation services available to children and adolescents with SCI in SIN unit catchment areas. In addition, telephone or Skype-interviews will be used to complement data when necessary.

The following main issues will be explored (detailed questionnaire is available):

I. Hospital setting, interaction with acute hospitals and referral processes II. Rehabilitation beds and patient case-mix III. Spinal rehabilitation and staffing and therapy intensity IV. Availability of secondary staff, ancillary services and support V. Life long follow-up

Also, the following background information will be collected:

1. SCI-prevention programmes in the region
2. Brief review of the implementation of child protection in each region

The questionnaire will be available both electronically and in a paper version in English and will be completed by the local principal investigator (PI) or by a representative from each of the participating units chosen by the local PI. The local PI will be a bilingual person with good local knowledge. Clarification of responses will occur in cooperation between the local PI and the project manager at Sunnaas. Descriptive analysis will be performed with the median and interquartile range (IQR) reported for numerical data not normally distributed.

Study II (explorative study/ interviews) An inductive, exploratory study with a qualitative design will be chosen to obtain a detailed description and understanding of how children aged of 13-17 years, perceive living with SCI in SIN-unit catchment areas.

Individual, face-to-face interviews will be conducted based on a thematic, semi-structured interview guide with relevant follow-up questions. The interviews will take place in the informant's home or another place chosen by the informant. Ninety minutes or more will be allowed for each interview. Due to Corona restrictions virual interviews on a safe digital platform like Teams or Norske Helsenett will be allowed. This apply especially for the additional Norwegian interviews as they are planned to take place during the autumn of 2020 and spring of 2021.

A semi-structured interview guide has been developed in cooperation between researchers and clinicians with experience in working with children and adolescents. Appropriate open ended questions are listed within each main area of the interview and key-questions are marked to assure that they are asked for. A salutogenic approach with strength based questions built on established principles and guidelines for psychosocial screening in young persons has been used (EuTEACH; HEEADSSS assessment; HEADSSS assessment, Clinical Practice Guidelines).

Themes in the semi-structured interview guide (detailed interview guide is available):

* The injury/ the accident
* Acute care, rehabilitation and follow-up
* Daily living with SCI with a pediatric onset
* Home, education/employment, eating, activities, drugs, sexuality, suicide/depression/self-image, safety (HEEADSSS)
* Resources and networks
* Health
* Peer learning/ role models
* The future/ life goals

Pilot interviews will be conducted to test the interview guide before deciding on a final version that will be translated to all relevant languages.

To assure that all interviews are conducted in a good manner in different units, an educational curriculum will be developed. Also, the interviewers will be trained in a 2-day seminar. All interviews will be taped with a digital voice recorder and transcribed verbatim in each unit. The transcripts will be translated to Norwegian by bilingual translators with knowledge of neurological rehabilitation and analyzed using inductive qualitative content analysis seeking to identify both manifest categories and underlying, latent meanings.

ETHICAL CONSIDERATIONS Ethical approval will be applied for in each country (Norway, Sweden, China, Russia, US, Israel and Palestine). All encoded material will be entered in a database at the Department of Research, Sunnaas Rehabilitation Hospital. Passkey will be stored separately and locked in a fireproof safe. Recorded/taped interviews will be transcribed and encoded and both the audio file (also encoded) and the transcript will be stored in a locked, fireproof safe.

Candidate participants will be approached and informed about the study by a letter. The letter will explain (1) the purpose of the study, (2) the procedures and (3) confidentiality. The participant will be informed about their right to withdraw at any time and for any reason without affecting your treatment by any means. The letter will include an 'Informed Consent Form' that he/she and his/her caregivers must sign and date and return to their study site before they can participate.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents (< 18 years)
* Diagnoses: either a non-traumatic or traumatic SCI after the age of 7
* Has been discharged from acute treatment phase for 6 months or more

Exclusion Criteria:

• Diagnosis of severe neurological conditions affecting the cognition of the child or adolescent (e.g. as a result of encephalocele or acquired brain injury)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents between the age of 13-17 years of age diagnosed with a non-traumatic or a traumatic SCI after the age 7.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Perception of psychosocial aspects | October 2018 - June 2021
  Qualitative individual indepth interviews
Organization and delivery of rehabilitation services | October 2018 - December 2020
  Web survey

SECONDARY OUTCOMES:
Translation and cross-cultural adaptation of PEDI SCI in to Norwegian | October 2020 - December 2022
  PEDI SCI

CONTACTS AND LOCATIONS:
Overall Officials: Johan K Stanghelle, Professor, Study Director — Sunnaas Rehabilitation Hospital, University of Oslo; Kirsti S Roaldsen, Professor, Principal Investigator — Sunnaas Rehab Hospital, Karolinska Institutet and Oslo Met
Locations (11):
- Rusk Institute of Rehabilitation Medicine, New York, New York, United States
- Peter New, Caulfield, Australia
- China (2):
  - China Rehabilitation and Research Center (CRRC), Beijing, Feng Tai District
  - No 81 Rehabilitation Center, Chengdu, Sichuan
- The Edmond & Lily Safra Children's Hospital, the Chaim Sheba Medical Center, Tel Aviv, Tel HaShomer, Israel
- Björneveien 11, Oslo, Bjørnemyr, Norway
- Bethlehem Arab Society of Specialized Rehabilitation and Surgery Hospital, Bethlehem, Palestinian Territories
- Policlinica 2 & Petrozavodsk City Children's Hospital, Petrozavodsk, Republic of Karelia, Russia
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Rehab Station Stockholm/ Spinalis, Solna

IPD SHARING:
Plan to Share IPD: No